CLINICAL TRIAL: NCT00214903
Title: European Active Surveillance Study of Women Taking HRT
Brief Title: European Active Surveillance Study of Women Taking Hormone Replacement Therapy (HRT)
Status: Completed | Type: Observational
Sponsor: Center for Epidemiology and Health Research, Germany (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Juergen Dinger, MD, PhD, Principal Investigator, Center for Epidemiology and Health Research, Germany
Other Study IDs: ZEG 2000_3
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Results first posted 2014-11-14 (Estimated); Last update posted 2014-12-01 (Estimated); Status verified 2014-11

CONDITIONS: Menopausal Symptoms
Keywords: Postmenopause; HRT

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: New users of oral continuous combined HRT containing drospirenone
- 2: New users of oral continuous combined HRT containing other progestagens

SUMMARY:
The objective of the active surveillance study is to compare incidence rates of serious adverse events in users of all types of newly prescribed oral continuous combined HRT products. The primary focus is the assessment of pertinent cardiovascular outcomes (such as venous and arterial thromboembolism) in new HRT users for up to 8.5 years.

DETAILED DESCRIPTION:
The safety of a novel drug product containing a new chemical entity should be assessed in an extensive post marketing safety surveillance program. It is also prudent to assess both, the safety outcomes that relate specifically to the targeted population, as well as those that could potentially be related to the special pharmacological characteristics of the novel drug product. Differentiating between the inherent background population risk and a potential incremental risk due to treatment is often challenging. Active safety surveillance using valid epidemiological study designs has been proven to be a pertinent and reliable method to approach this endeavour.

The primary objective of the study, the European Active Surveillance Study of Women taking HRT (EURAS-HRT), is to compare incidence rates of serious adverse events in users of all types of newly prescribed oral continuous combined HRT products. This active surveillance study will assess pertinent cardiovascular outcomes in new HRT users over a study period of up to 8.5 years. Also, all other serious adverse events will be reported.

The new drug product under surveillance in the EURAS - HRT study contains the novel synthetic progestagen drospirenone (DRSP) combined with estradiol.

As estrogen/progestagen combinations increase the risk for thromboembolism, all new drug products that contain a novel estrogen or progestagen should be investigated for their influence on venous and arterial thromboembolic events rates. A large, prospective, controlled cohort study of OC users (EURAS OC study), which compared DRSP-containing OC users with other OC users, demonstrated that DRSP is not associated with an increased incidence for any of the above-mentioned adverse events in OC users. However, because OC users are two to three decades younger than the typical HRT user the results of the OC study can only partially be extrapolated to older age groups.

The participating women will complete a baseline survey using a self-administered questionnaire to describe the baseline risk. After 6 months, 12 months, and then on an annual basis, they will fill out a questionnaire in which they record complaints and events during the use of the prescribed HRTs. All adverse outcomes (including cancer) occurring during the observational period will be evaluated additionally. Reported serious adverse events will be validated and analyzed. As study participants may switch from oral continuous combined products to other oral or non-oral HRT products the outcomes for these preparation are recorded too. However, these results represent not the scientific focus of the study.

Based on experience obtained in previous HRT studies, complex sources of bias and confounding are expected. Multivariate methods will therefore be used to adjust for confounding.

ELIGIBILITY:
Inclusion Criteria:

* All women aged 40 or more years who started use of a new oral HRT at the time of inclusion in the study

Exclusion Criteria:

* Women who do not consent to participate in the study

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women aged 40 or more years using HRT
Sampling Method: Non-Probability Sample
Enrollment: 30597 (Actual)
Dates: Start 2004-11; Primary Completion 2011-05 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Dinger, MD, PhD, Principal Investigator — ZEG, Invalidenstrasse 115, 10115 Berlin, Germany
Locations (1):
- Center for Epidemiology and Health Research, Berlin, Germany

REFERENCES:
- [Derived] Dinger J, Bardenheuer K, Heinemann K. Drospirenone plus estradiol and the risk of serious cardiovascular events in postmenopausal women. Climacteric. 2016 Aug;19(4):349-56. doi: 10.1080/13697137.2016.1183624. Epub 2016 May 13. PMID 27174159

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 31,321 patients were recruited for the EURAS HRT study. 724 patients were excluded due to protocol violations (e.g., patient agreed to participate but never started to use the new HRT preparation or continued to use a previously prescribed preparation).
Groups:
- DRSP/E2: Users of oral continuous combined preparations containing 2mg DRSP and 1mg estradiol
- ooccHRT: Users of other oral continuous combined HRT preparations containing other progestogens
- ooHRT: Users of oral but not continuous combined HRT preparations
- Non-oral HRT: Users of non-oral HRT preparations
Period: Overall Study
Arm/Group | DRSP/E2 | ooccHRT | ooHRT | Non-oral HRT
Started | 10043 | 13384 | 4113 | 3057
Completed | 10043 | 13384 | 4113 | 3057
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: At baseline, 33% of women were using DRSP/E2, 44% were using ooccHRT, 13% were using ooHRT, and 10% 'Non-oral HRT'. These proportions only partially reflect the overall exposure in each cohort (AT population) because market authorization for DRSP/E2 was delayed by more than 1.5 years.
Groups:
- Total: Total of all reporting groups
Arm/Group | DRSP/E2 | ooccHRT | ooHRT | Non-oral HRT | Total
Number analyzed (Participants) | 10043 | 13384 | 4113 | 3057 | 30597
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (6.4) | 55.1 (6.9) | 52.9 (8.3) | 56.2 (7.7) | 54.0 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10043 | 13384 | 4113 | 3057 | 30597
  Male | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — This study was conducted in seven European countries: Austria, Belgium, Germany, Italy, the Netherlands, Spain, and Turkey. 23,025 participants were eligibly enrolled in Central Europe, and 7,572 participants in Southern Europe.
  participants
    Europe | 10043 | 13384 | 4113 | 3057 | 30597

OUTCOME MEASURES:

1. Primary Outcome: Venous Thromboembolism (e.g., Deep Venous Thrombosis and Pulmonary Embolism)
Description: Venous thromboembolism (VTE) linked to the use of continuous combined HRT containing both drospirenone (DRSP) and estradiol (E2) or to other oral continuous combined HRT preparations.
Time Frame: within 8.5 years
Population: The number of participants refers to the ITT study population. During the course of the study, women could for example stop hormonal treatment at any point of time. Therefore, the woman-years of exposure for each group are provided in addition.
Measure: Number; unit: participants
Units Other Than Participants: Women-years
Arm/Group | DRSP/E2 | ooccHRT | ooHRT | Non-oral HRT
Number analyzed (Participants) | 10043 | 13384 | 4113 | 3057
Number analyzed (Women-years) | 13,714 | 31,938 | 9,253 | 7,785
participants | 24 | 74 | 21 | 12
Statistical Analysis 1: Comparison: DRSP/E2 vs ooccHRT; Tested null hypotheses: the VTE hazard ratio for DRSP/E2 vs. ooccHRT is higher or equal to 2; Test type: Non-Inferiority or Equivalence — Sample size calculations were based on a non-inferiority test to exclude a two-fold risk of cardiovascular events in users of DRSP/E2 compared to other oral continuous combined HRT. These calculations are based on the following assumptions: 1) one-sided α 0.05; 2) power (1-β) of 0.80; 3) Estimated incidence of cardiovascular events, ATE and VTE would be at least 1.0, 0.3 and 0.2 event/100 woman-years and 4) non-inferiority limit hazard ratio of 2; Hazard Ratio (HR) = 0.8, 95% CI 2-sided [0.5 to 1.3] — Hazard ratio was adjusted for age, BMI, duration of current use, family history of VTE, region, and HRT user status

2. Primary Outcome: Arterial Thromboembolism (e.g., Acute Myocardial Infarction and Stroke)
Description: Arterial thromboembolism (ATE) linked to the use of continuous combined HRT containing both drospirenone (DRSP) and estradiol (E2) or to other oral continuous combined HRT preparations.
Time Frame: within 8.5 years
Population: as for outcome 1
Measure: Number; unit: participants
Units Other Than Participants: Women-years
Arm/Group | DRSP/E2 | ooccHRT | ooHRT | Non-oral HRT
Number analyzed (Participants) | 10043 | 13384 | 4113 | 3057
Number analyzed (Women-years) | 13,714 | 31,938 | 9,253 | 7,785
participants | 15 | 95 | 33 | 23
Statistical Analysis 1: Comparison: DRSP/E2 vs ooccHRT; Tested null hypotheses: the ATE hazard ratio for DRSP/E2 vs. ooccHRT is higher or equal to 2; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.5, 95% CI 2-sided [0.3 to 0.8] — Hazard ratio was adjusted for age, BMI, hypertension, diabetes, family history of fatal ATE, region, and smoking

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected over a time period of 8.5 years.
Description: Complete cohorts, as-treated population. All study participants were asked for adverse events at each follow-up.
Arm/Group | DRSP/E2 | ooccHRT | ooHRT | Non-oral HRT
Serious Adverse Events (participants affected / at risk) | 707/10043 | 1998/13384 | 576/4113 | 508/3057
Other Adverse Events (participants affected / at risk) | 0/10043 | 0/13384 | 0/4113 | 0/3057
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DRSP/E2 (N=10043) | ooccHRT (N=13384) | ooHRT (N=4113) | Non-oral HRT (N=3057)
Infectious diseases (Infections and infestations) | 12 (12) | 28 (28) | 8 (8) | 9 (9) — Prespecified category; a further breakdown by sub-categories was only planned in case that the results indicated an increased risk for DRSP/E2.
Neoplasms, malignant and benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 91 (91) | 248 (248) | 62 (62) | 58 (58) — Prespecified category; a further breakdown by sub-categories was only planned in case that the results indicated an increased risk for DRSP/E2.
Diseases of the blood and bloodforming organs (Blood and lymphatic system disorders) | 1 (1) | 7 (7) | 2 (2) | 1 (1) — Prespecified category; a further breakdown by sub-categories was only planned in case that the results indicated an increased risk for DRSP/E2.
Endocrine diseases (Endocrine disorders) | 11 (11) | 36 (36) | 8 (8) | 8 (8) — Prespecified category; a further breakdown by sub-categories was only planned in case that the results indicated an increased risk for DRSP/E2.
Psychiatric and neurological disorders (Psychiatric disorders) | 50 (50) | 112 (112) | 33 (33) | 32 (32) — Prespecified category; a further breakdown by sub-categories was only planned in case that the results indicated an increased risk for DRSP/E2.
Eye (Eye disorders) | 13 (13) | 32 (32) | 12 (12) | 10 (10) — Prespecified category; a further breakdown by sub-categories was only planned in case that the results indicated an increased risk for DRSP/E2.
Ear (Ear and labyrinth disorders) | 14 (14) | 32 (32) | 9 (9) | 7 (7) — Prespecified category; a further breakdown by sub-categories was only planned in case that the results indicated an increased risk for DRSP/E2.
Cardiovascular system (Cardiac disorders) | 135 (135) | 542 (542) | 155 (155) | 130 (130) — Prespecified category; a further breakdown by sub-categories was only planned in case that the results indicated an increased risk for DRSP/E2.
Respiratory system (Respiratory, thoracic and mediastinal disorders) | 33 (33) | 78 (78) | 27 (27) | 22 (22) — Prespecified category; a further breakdown by sub-categories was only planned in case that the results indicated an increased risk for DRSP/E2.
Digestive system (Gastrointestinal disorders) | 90 (90) | 237 (237) | 69 (69) | 68 (68) — Prespecified category; a further breakdown by sub-categories was only planned in case that the results indicated an increased risk for DRSP/E2.
Skin (Skin and subcutaneous tissue disorders) | 7 (7) | 24 (24) | 5 (5) | 5 (5) — Prespecified category; a further breakdown by sub-categories was only planned in case that the results indicated an increased risk for DRSP/E2.
Muscoskeletal system & connective tissue (Musculoskeletal and connective tissue disorders) | 117 (117) | 285 (285) | 85 (85) | 70 (70) — Prespecified category; a further breakdown by sub-categories was only planned in case that the results indicated an increased risk for DRSP/E2.
Genitourinary system (Reproductive system and breast disorders) | 40 (40) | 111 (111) | 29 (29) | 24 (24) — This adverse event term also includes renal and urinary disorders. Prespecified category; a further breakdown by sub-categories was only planned in case that the results indicated an increased risk for DRSP/E2.
Injury, poisoning, accidents, etc. (Injury, poisoning and procedural complications) | 93 (93) | 226 (226) | 72 (72) | 64 (64) — Prespecified category; a further breakdown by sub-categories was only planned in case that the results indicated an increased risk for DRSP/E2.

LIMITATIONS AND CAVEATS:
In non-experimental studies like EURAS-HRT the possibility of bias and residual confounding can never be entirely eliminated. The findings may exclude large, but not small relative risks.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes